CLINICAL TRIAL: NCT05371769
Title: Evaluation of the Efficiency of the Chronic Pain Management Education Program Developed for Nursing Students
Brief Title: Evaluation of the Efficiency of the Chronic Pain Management Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nefise Cevriye SUCU ÇAKMAK, Principal Investigator, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NSUCUCAKMAK
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Nursing Caries; Chronic Pain
Keywords: Chronic pain; Nursing student education; Web-Technology based education
MeSH Terms: conditions — Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomization: After applying the exclusion criteria to a total of 94 students, the students who accepted to participate in the study was randomly selected into two groups (A and B) of 35 students by simple random sampling by creating a computer-assisted simple random numbers table (www.randomizer.org). Selected students was randomly assigned so that the general academic achievement grades of both groups were homogeneous. The groups was randomly assigned to the intervention or control group by the code "A" and "B" by the software specialist.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It was explained to all students that training was given over the website https://www.agriegitimi.net and the starting time of the training was announced on the website. Students were told that they were be able to attend training and testing at the relevant time according to notifications. Students were not know that they were in the experimental or control group. In this way, students were blinded. Only the software specialist could know the students in the intervention and control groups. The data could sent to the statistician by the software specialist as group A and B data. This way the statistician could be blind. The researcher could not present at any stage of data collection. After the statistical analysis was done and the research report was written, the coding of the experimental and control groups were explained to the researcher by the software specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): The students in the control group will be given a pre-test, and two weeks later, the post-test will be applied. After the chronic pain education group completes the research, the chronic pain education program will be opened to the students in the control group, too.
  Interventions: Other: No intervention
- Chronic pain education group (Experimental): The pre-test will be opened to the students in the chronic pain education group simultaneously with the opening of the post-tests for the control group.After the students in the chronic pain education group completed the pre-test, the chronic pain management training program developed for nursing students will be applied for 2 weeks. Post test will be applied at the end of all training videos and evaluation questions.
  Interventions: Other: chronic pain management education program

INTERVENTIONS:
Other: chronic pain management education program — The chronic pain management training program will be applied for 2 weeks. The training consists of 15 videos about theory and practice topics in chronic pain management. There are evaluation questions at the end of each video.
  Other Names: Experimental group
  Arms: Chronic pain education group
Other: No intervention — No intervention will be made.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The research will be conducted to evaluate the effectiveness of the web-based chronic pain management training program developed for nursing students. It is planned in a randomized controlled triple-blind design with the final year nursing students of the Nursing Department of Çankırı Karatekin University in a pre-test-post-test order.

ELIGIBILITY:
Inclusion Criteria:

* Nursing Grade 4
* with internet access
* Students who volunteered to participate in the research

Exclusion Criteria:

* Having a diagnosed psychiatric disorder
* Difficulty in understanding and speaking Turkish
* Graduated from Health Vocational High School
* Attending any training on pain and/or having a pain education certificate

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Introductory features form | pre-intervention
  It was prepared by the researcher in line with the literature knowledge. In the form of introductory characteristics of nursing students; There are 7 questions about the students' date of birth, gender, whether they have chronic pain, whether they have chronic pain from family members they live with, in which clinics they do internship, and whether they find themselves competent in the management of chronic pain of the patients they care for.
Scale of attitudes of students studying in the field of health towards patients with chronic pain | pre-intervention
  The Attitude Scale of Health Students towards Patients with Chronic Pain is a 5-point Likert scale and has 18 items. It consists of two factors: sensitivity orientation and error orientation. The Cronbach's Alpha coefficients are 0.88 and 0.75 for the first and second factors, respectively. Each factor gets a separate score. Each item in the factors receives a score between "1" and "5". The scores are summed up and divided by the number of items, then a score between 1 and 5 is obtained, thus a standard evaluation of two factors can be done. There is no cut-off score in the scale.
  An increased score from the sensitivity and misconception orientation factors indicates that healthcare professionals' attitude towards patients with chronic pain is positively strong. On the other hand, a low score on these factors indicates a strong negative attitude.
Scale of attitudes of students studying in the field of health towards patients with chronic pain | immediately after the intervention
  The Attitude Scale of Health Students towards Patients with Chronic Pain is a 5-point Likert scale and has 18 items. It consists of two factors: sensitivity orientation and error orientation. The Cronbach's Alpha coefficients are 0.88 and 0.75 for the first and second factors, respectively. Each factor gets a separate score. Each item in the factors receives a score between "1" and "5". The scores are summed up and divided by the number of items, then a score between 1 and 5 is obtained, thus a standard evaluation of two factors can be done. There is no cut-off score in the scale.
  An increased score from the sensitivity and misconception orientation factors indicates that healthcare professionals' attitude towards patients with chronic pain is positively strong. On the other hand, a low score on these factors indicates a strong negative attitude.
Chronic pain management knowledge test | pre-intervention
  The knowledge test on chronic pain management was created by the researchers in line with the literature. The knowledge test for chronic pain management includes 24 case-based five-choice multiple-choice questions. In this test, each correct answer is 1 point and a wrong answer is zero. The total score is obtained by adding the scores obtained from the test. The highest score that can be obtained from the test is 24, and the lowest score is zero. An increase in the score obtained from the test indicates that the participant's level of knowledge about chronic pain management increases, while a decrease in the score indicates a low level of knowledge.
Chronic pain management knowledge test | immediately after the intervention
  The knowledge test on chronic pain management was created by the researchers in line with the literature. The knowledge test for chronic pain management includes 24 case-based five-choice multiple-choice questions. In this test, each correct answer is 1 point and a wrong answer is zero. The total score is obtained by adding the scores obtained from the test. The highest score that can be obtained from the test is 24, and the lowest score is zero. An increase in the score obtained from the test indicates that the participant's level of knowledge about chronic pain management increases, while a decrease in the score indicates a low level of knowledge.
Chronic pain management training program evaluation form | immediately after the intervention
  Chronic pain management training program evaluation Form, Game-based virtual reality application evaluation form in Bıyık-Bayram and Çalışkan's (2017) The Effects of Game-Based Virtual Reality Application on Nursing Students' Learning Tracheostomy Care, was revised and revised to the chronic pain management training program. has been prepared. This form consists of two parts. The first part consists of two open-ended questions about the positive and negative thoughts of the students about the chronic pain management education program, and the second part consists of 16 questions that include 5-point Likert-type scoring in which the statements about the education program are evaluated. Each item in the form receives a score between "1" and "5". An increase in the score obtained from the form indicates that the participant evaluated the chronic pain management training program p vely.This form will be filled by the students in the experimental group at the end of the post-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Cevriye SUCU ÇAKMAK, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No